CLINICAL TRIAL: NCT00595322
Title: Safety of Bevacizumab in the Radiation Treatment of Recurrent Malignant Glioma: A Pilot Study
Brief Title: Bevacizumab in the Radiation Treatment of Recurrent Malignant Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-092
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Brain Cancer; Recurrent Malignant Gliomas; Primary Brain Tumor
Keywords: Bevacizumab; Radiation Treatment; Brain Cancer
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Bevacizumab; Radiation

ARMS (1):
- 1 (Experimental): bevacizumab and radiation (IMRT)
  Interventions: Other: bevacizumab and radiation (IMRT)

INTERVENTIONS:
Other: bevacizumab and radiation (IMRT) — bevacizumab 10 mg/kg IV once every two weeks on days 1 and 15 of every cycle (cycle defined as 28 days). If the tumor volume remains < 40 cc, the patient will undergo stereotactic radiotherapy with IMRT (30Gy) beginning anywhere from day 7-10 of cycle 2 (5 doses of 6 Gy over 2 and a half weeks)

SUMMARY:
This is a pilot study. The goal of this study is to test whether Bevacizumab is safe enough in patients with brain tumors so that a larger study can be conducted. This study will also give us some information about whether the combination of Bevacizumab and radiation has potential to become an effective treatment for regrowing brain tumors.

Bevacizumab is an experimental drug that blocks a molecule called VEGF that is found in high amounts in malignant gliomas. VEGF promotes the growth of blood vessels that bring nutrients to tumor cells. In studies with laboratory animals, Bevacizumab slowed the growth of several different types of human cancer cells by blocking the effects of VEGF. There is also evidence that Bevacizumab enhances the effects of radiation on tumor cell

ELIGIBILITY:
Inclusion Criteria:

* Recurrent malignant glioma that has failed prior radiotherapy and/or chemotherapy. Surgery for the recurrence may be offered to selected patients prior to receiving bevacizumab and IMRT on this protocol.
* MRI scan with gadolinium contrast showing geographically-circumscribed tumor < than or equal to 3.5cm. (Scan must be performed on a steroid dosage that has been stable for at least 5 days. If the steroid dose is increased between date of imaging and registration, a new baseline MRI is required).
* Patients must have recovered from the toxic effects of prior therapy:
* An interval of > than or equal to 4 weeks (28 days) from prior cytotoxic therapy
* An interval of > than or equal to 1 week (7 days) from any non-cytotoxic agents
* An interval of > than or equal to 6 weeks (42 days) from the completion of radiation therapy
* Absolute neutrophil count > than or equal to 1,500/mm3.
* Platelet count > than or equal to 100,000/mm3.
* Hemoglobin > than or equal to 10 g/dl.
* BUN and serum creatinine both < 1.5 times upper limit of normal.
* Total bilirubin both < 1.5 times upper limit of normal.
* SGOT and SGPT both < than or equal to 3 times upper limit of normal.
* Alkaline phosphatase < than or equal to 2 times upper limit of normal.
* > than or equal to 18 years of age.
* Karnofsky Performance Score > or equal to 70
* Life expectancy > or equal to 12 weeks
* Men and women with reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.
* Patient or their legal proxy must provide written informed consent prior to registration on study.

Exclusion Criteria:

* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study.
* Blood pressure >150 mmHg systolic and/or >100 mmHg diastolic
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* Unstable angina within 12 months of study enrollment
* CTC 3.0 Grade 2 or greater congestive heart failure
* History of myocardial infarction within 12 months of study enrollment
* History of stroke or transient ischemic attack at any time
* Known CNS disease
* Known hypersensitivity to any component of bevacizumab
* History of peptic ulcer within the last 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Use of ongoing anticoagulants or antiplatelet agents (aspirin, NSAIDS, etc)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the first dose of bevacizumab or anticipation of need for major surgical procedure during the course of the study. (Recently resected patients may be enrolled on-study two weeks post-surgery. However, treatment with Bevacizumab will not begin until 28 days after the surgical procedure for all patients.)
* Craniotomy wound that has not sufficiently healed
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to study enrollment
* Pregnant (positive pregnancy test) or lactating
* Urine protein:creatinine ratio ≥1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Lung carcinoma of squamous cell histology or any histology in close proximity to a major vessel, cavitation, or history of hemoptysis
* Inability to comply with study and/or follow-up procedures
* Glioma showing prior spontaneous hemorrhage as determined from the clinical history or from any preoperative CT or MRI scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
To test the safety of bevacizumab in patients with recurrent malignant gliomas in preparation for a larger study to test the efficacy of this drug used during the initial radiation treatment of these tumors if safety is affirmed. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gutin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Gutin PH, Iwamoto FM, Beal K, Mohile NA, Karimi S, Hou BL, Lymberis S, Yamada Y, Chang J, Abrey LE. Safety and efficacy of bevacizumab with hypofractionated stereotactic irradiation for recurrent malignant gliomas. Int J Radiat Oncol Biol Phys. 2009 Sep 1;75(1):156-63. doi: 10.1016/j.ijrobp.2008.10.043. Epub 2009 Jan 23. PMID 19167838
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org